CLINICAL TRIAL: NCT06570122
Title: Effectiveness of AI-powered Mobile Phone-based Interventions in Parental Smoking Cessation
Brief Title: Mobile Phone-Based Smoking-Cessation Intervention for Smoking Parents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mCessation in smoking parents
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI chatbot support group (Experimental): AI-powered chatbot support+ 5A's/5R's advice + health warning leaflet
  Interventions: Behavioral: 5A's/5R's advice; Other: Health warning leaflet; Behavioral: AI-powered chatbot support
- Control group (Active Comparator): 5A's/5R's advice + health warning leaflet
  Interventions: Behavioral: 5A's/5R's advice; Other: Health warning leaflet

INTERVENTIONS:
Behavioral: 5A's/5R's advice — 5A's (Ask, Advise, Assess, Assist, Arrange) for smokers who are ready to quit, and 5R's (relevance, risks, rewards, roadblocks, and repetition) for smokers who are not ready to quit.
Other: Health warning leaflet — The health warning leaflet provides essential information on the dangers of secondhand and thirdhand smoke. It outlines how exposure to these forms of smoke can harm both smokers and non-smokers, particularly children, by increasing the risk of respiratory illnesses and other health issues.
Behavioral: AI-powered chatbot support — Participants will receive three months of AI-powered chatbot, equipped with personalized interactions and real-time support, via WeChat.
  Arms: AI chatbot support group

SUMMARY:
This study aims to explore the feasibility and preliminary effectiveness of a mobile phone-based intervention tailored specifically for smoking parents.

DETAILED DESCRIPTION:
Parental smoking is associated with numerous adverse outcomes, including exposure to secondhand smoke, heightened risk of respiratory illnesses in children, and an increased likelihood that children will adopt smoking behaviors themselves. Despite awareness of these risks, many parents find it challenging to quit smoking due to stress, lack of support, and time constraints.

This randomized controlled trial (RCT) investigates the effectiveness of a mobile phone-based intervention tailored specifically for smoking parents. The intervention group will receive AI-powered chatbot cessation support, while the control group will be provided with brief cessation advice. The study aims to determine whether the AI-driven intervention is more effective in helping parents quit smoking compared to traditional brief advice.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and above, reside in Zhuhai for the next 6 months
2. smoke at least 1 cigarette or use e-cigarettes daily
3. have a smartphone and a WeChat account, able to use WeChat skillfully

Exclusion Criteria:

1. Smokers who have communication barrier (either physically or cognitively)
2. Smokers who are currently participating in other SC programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 3 and 6 months follow-up
  Self-reported 7-day point prevalence quit rate in the two groups
Eligibility rate | baseline
  the percentage of eligible smokers out of the total number of smokers screened

SECONDARY OUTCOMES:
Consent rate | baseline
  the percentage of eligible smokers who agree to participate out of the total number of eligible smokers
Percentage of Participant Engagement with E-Messages and Counselor Chats | 3 months follow-up
  This outcome measures the percentage of participants who engage with the intervention by reading e-messages and responding to counselor chat messages at least once during the 3-month follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No